CLINICAL TRIAL: NCT00831090
Title: Endothelial Function and Vein Graft Remodeling
Acronym: EFVGR
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-02338; HL92163-01
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Peripheral Arterial Disease; Cardiovascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A segment of vein that would usually be discarded will be taken to a lab for testing of endothelial reactivity and quantification of endothelial coverage through CD31 staining.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to better understand why some vein bypass grafts develop narrowing. Evidence suggests that there is a relationship between inflammatory markers in the blood and the narrowing that occurs in blood vessels. In this study, we will look at inflammatory markers in the blood and how well the vein graft functions.

DETAILED DESCRIPTION:
Despite the acceptance of catheter-based approaches to lower extremity reconstruction, bypass with autogenous vein remains the most durable option. In the United States alone there are approximately 100,000 lower extremity bypass procedures performed yearly. However, 30-50% of these grafts either occlude or require revision in the first 5 years.

Traditional Framingham cardiovascular risk factors such as dyslipidemia and diabetes do not predict which grafts are at risk for failure. Therefore other variables such as hemodynamic factors or endothelial function may be important in identifying vulnerable vein grafts. The applicant has previously noted that vein grafts undergo dramatic geometric remodeling within the first month after implantation into the arterial circulation. This is partly driven by hemodynamic forces such as shear stress and is thought to be related to endothelial function. Shear stress is positively correlated with early (0-1 month) luminal enlargement. This adaptive response is important to maintain bypass graft patency. However, there is considerable amount of variability in this response unaccounted for by shear stress alone. The applicant has further shown that baseline systemic inflammation dampens the ability for adequate vein graft luminal expansion and therefore may uncouple the mechano-chemical signal transduction at the endothelial level. Therefore, this study will examine the relationship between circulating levels of inflammatory mediators and endothelial function in a cohort of patients undergoing lower extremity arterial reconstruction with autogenous vein.

ELIGIBILITY:
Inclusion Criteria:

* Age > 22 or < 90 years
* Undergoing lower extremity (infrainguinal) bypass using autologous vein for the treatment of disabling claudication or critical limb ischemia secondary to chronic atherosclerotic occlusive disease
* Able to understand, give, and take part in the consent process

Exclusion Criteria:

* Age < 22 or > 90 years
* Grafts employing prosthetic or other non-autologous vein material in any part (e.g. composite grafts). [Patch angioplasty of inflow and outflow vessel permissible with any material]
* Vasculitis, trauma, acute embolic disease as etiology of limb ischemia
* History of diagnosed hypercoagulable state
* Evidence of active infection - pneumonia, urinary tract, etc., requiring medical therapy
* Evidence of significant local sepsis in foot or limb prior to bypass
* Patients taking immunosuppressant medications (steroids, chemotherapeutic agents)
* Other concurrent significant illness within 30 days
* Non-English speakers

Ages: 22 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vascular Surgery clinic
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-01; Primary Completion 2015-01-16 (Actual); Study Completion 2015-01-16 (Actual)

PRIMARY OUTCOMES:
Successful early vein graft remodeling | 3 Months
  An increase in vein graft lumen diameter at three months

CONTACTS AND LOCATIONS:
Overall Officials: Warren J. Gasper, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California